CLINICAL TRIAL: NCT04918511
Title: An Open-label Phase I, Dose Escalation Study of the Safety and Tolerability of OPD5 as Myeloablative Conditioning Regimen Followed by Autologous Stem Cell Transplant (ASCT) for Patients With Relapsed Refractory Multiple Myeloma (RRMM)
Brief Title: A Study of OPD5 Followed by Autologous Stem Cell Transplant for Patients With Relapsed Refractory Multiple Myeloma
Acronym: COAST
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor made the decision to terminate the COAST study to refocus the OPD5 clinical program.
Sponsor: Oncopeptides AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OP-501
Record Dates: First submitted 2021-05-27; First posted 2021-06-09 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Relapse Multiple Myeloma; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: A minimum of 3 and up to 6 evaluable patients will be enrolled per dose level. After the first cohort, the doses for the following dose cohorts will be adaptively escalated/de-escalated based on observed dose limiting toxicities in previous cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Dose cohort 1 (Experimental): In dose cohort 1, treatment with OPD5 solution will be given as one single i.v. infusion over 30 minutes at a dose level of 30 mg/m2 (dose based on body surface area)
  Interventions: Drug: OPD5
- Dose cohort 2 (Experimental): In dose cohort 2, treatment with OPD5 solution will be given as one single i.v. infusion over 30 minutes at a dose level decided based on the results from Dose Cohort 1
  Interventions: Drug: OPD5
- Dose cohort 3 (Experimental): In dose cohort 3, treatment with OPD5 solution will be given as one single i.v. infusion over 30 minutes at a dose level decided based on the results from Dose Cohort 2
  Interventions: Drug: OPD5
- Dose cohort 4 (Experimental): In dose cohort 4, treatment with OPD5 solution will be given as one single i.v. infusion over 30 minutes at a dose level decided based on the results from Dose Cohort 3
  Interventions: Drug: OPD5
- Dose cohort 5 (Experimental): In dose cohort 5, treatment with OPD5 solution will be given as one single i.v. infusion over 30 minutes at a dose level decided based on the results from Dose Cohort 4
  Interventions: Drug: OPD5
- Dose cohort 6 (Experimental): In dose cohort 6, treatment with OPD5 solution will be given as one single i.v. infusion over 30 minutes at a dose level decided based on the results from Dose Cohort 5
  Interventions: Drug: OPD5
- Dose cohort 7 (Experimental): In dose cohort 7, treatment with OPD5 solution will be given as one single i.v. infusion over 30 minutes at a dose level decided based on the results from Dose Cohort 6
  Interventions: Drug: OPD5

INTERVENTIONS:
Drug: OPD5 — OPD5 solution for i.v. infusion

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of a single infusion of OPD5 before Autologous Stem Cell Transplant in patients with RRMM. The study will evaluate increasing doses of OPD5 to find the best dose and to assess any side effects. Each patient will be assigned to a dose cohort of 3-6 patients to receive one single dose of OPD5. Each patient will be hospitalized for about 14 days from the OPD5 infusion and then have monthly visits to the clinic for 3 months and then every third month until disease progression or starting new myeloma treatment, maximum up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between the ages of 18 years and 70 years at the planned time of study treatment; patients greater than 70 years of age may qualify on a case by case basis
* Diagnosis of multiple myeloma
* Received a previous Autologous Stem Cell Transplantation ( ASCT) (single or tandem) that resulted in disease progression within 24 months
* Received at least 2 prior lines of therapy
* Refractory to previous treatment with a Proteasome Inhibitor (PI), an immunomodulatory drug (IMiD) and an anti-Cluster of Differentiation 38 monoclonal antibody (anti-CD38 mAb)
* Male and women of childbearing potential agrees to use contraception during the treatment period and during a specified time period after the last dose

Exclusion Criteria:

* Prior treatment with melphalan flufenamide (melflufen) or OPD5
* Any medical condition that may interfere with safety or participation in this study
* Other malignancy diagnosed or requiring treatment within the past 3 years with the exception of adequately treated basal cell carcinoma, squamous cell skin cancer, carcinoma in-situ of the cervix or breast or very low and low risk prostate cancer in active surveillance
* Prior allogeneic stem cell transplantation or prior salvage ASCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-27 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and grade of Treatment Emergent Adverse Events (TEAEs) | 30 days post OPD5 treatment with ASCT
  Including frequency and grade of defined Dose Limiting Toxicities
Incidence of clinically significant changes in clinical laboratory parameters | 30 days post OPD5 treatment with ASCT
Magnitude of clinically significant changes in clinical laboratory parameters | 30 days post OPD5 treatment with ASCT
Incidence of clinically significant adverse findings in vital signs | 30 days post OPD5 treatment with ASCT
Severity of clinically significant adverse findings in vital signs | 30 days post OPD5 treatment with ASCT
Incidence of clinically significant adverse findings in electrocardiograms (ECGs) | 30 days post OPD5 treatment with ASCT
Severity of clinically significant adverse findings in electrocardiograms (ECGs) | 30 days post OPD5 treatment with ASCT
Incidence of clinically significant adverse findings in other physical examination parameters | 30 days post OPD5 treatment with ASCT
Severity of clinically significant adverse findings in other physical examination parameters | 30 days post OPD5 treatment with ASCT
Incidence of mucositis | 30 days post OPD5 treatment with ASCT
Severity of mucositis | 30 days post OPD5 treatment with ASCT
  Using World Health Organization (WHO) oral toxicity scale, from 0 (no change) to 4 (oral feeding is not possible)
The number of deaths not related to relapse or progression | 100 days post OPD5 treatment with ASCT

SECONDARY OUTCOMES:
Best Response | 30 days post OPD5 treatment with ASCT
  Best response for a single patient. Best response will include the following categories: stringent Complete Response (sCR), Complete Response (CR), Very Good Partial Response (VGPR), Partial Response (PR), Minimal Response (MR), Stable Disease (SD) and Progressive Disease (PD) as assessed by the investigator according to International Myeloma Working Group Uniform Response Criteria (IMWG-URC)
Overall Response Rate (ORR) | approximately 100 days post OPD5 treatment with ASCT
  Proportion of patients who achieve response of CR, sCR, VGPR or PR as their best response.
Duration of response (DOR) | approximately 12 months
  Time from the first confirmed response of sCR, CR, VGPR or PR to first confirmed disease progression, or death due to any cause
Time to progression (TTP) | approximately 12 months
  Time from the date of OPD5 administration to the date of the first documented confirmed PD
Time to next treatment (TTNT) | approximately 12 months
  Time from the date of OPD5 administration start to the start of first post study myeloma therapy (maintenance MM treatment not considered as new line of therapy)
Progression Free Survival (PFS) | approximately 12 months
  Time from the date of OPD5 dosing to the date of first documentation of confirmed progressive disease (PD) or death due to any cause
Pharmacokinetics Area under the curve AUC(0-t) for OPD5 and the metabolites desethyl-melflufen and melphalan | Day -1 (the day of OPD5 infusion)
Pharmacokinetics AUC(0-infinity) for OPD5 and the metabolites desethyl-melflufen and melphalan | Day -1 (the day of OPD5 infusion)
Pharmacokinetics elimination half-life (t½) for OPD5 and the metabolites desethyl-melflufen and melphalan | Day -1 (the day of OPD5 infusion)
Pharmacokinetics Cmax for OPD5 and the metabolites desethyl-melflufen and melphalan | Day -1 (the day of OPD5 infusion)
Time to hematological recovery | approximately Day 14
  defined as the return of Absolute Neutrophil Count (ANC) ≥ 0.5 x 10^9/L and platelets ≥ 20 x 10^9/L for two consecutive days
Time to myeloablation | approximately Day 14
  defined as the first of at least two consecutive days with ANC < 0.5 x 10^9/L and platelets <20 x 10^9/L
Minimal Residual Disease (MRD) status by Next Generation sequencing (NGS) in patients that achieve a CR or VGPR. | approximately Day 100

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Giralt, MD, Principal Investigator — Memorial Sloan Kettering Cancer Centre, New York City, United States
Locations (3):
- Czechia (3):
  - University Hospital Brno, Clinic of Internal Medicine - Hematology and Oncology, Brno
  - University Hospital Ostrava, Clinic of Hematooncology, Ostrava
  - Charles University and General Hospital in Prague, 1st Department of Medicine - Department of Hematology, First Faculty of Medicine, Prague